CLINICAL TRIAL: NCT04819282
Title: Use of Surgical Masks in the COVID-19 Pandemic: Does it Affect Physical Performance in Geriatrics?
Brief Title: Mask Usage and Physical Performance During COVID-19 Pandemic in Geriatrics
Status: Completed | Type: Observational
Sponsor: KTO Karatay University (Other)
Responsible Party: Principal Investigator, Büşra Alkan, Lecturer, KTO Karatay University
Other Study IDs: KaratayU4
Record Dates: First submitted 2021-03-24; First posted 2021-03-26 (Actual); Last update posted 2021-04-01 (Actual); Status verified 2021-03

CONDITIONS: Exercise Capacity; Geriatric; Mask
Keywords: Mask Usage; Geriatrics; Exercise Capacity; Physical Performance; Senior Fitness Test

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Week
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- One group: Physical performance was evaluated with the Senior Fitness Test in one group of geriatric individuals.
  Interventions: Diagnostic Test: Senior Fitness Test

INTERVENTIONS:
Diagnostic Test: Senior Fitness Test — Senior Fitness Test, simple and easy to use, was used to evaluate physical performance.

SUMMARY:
In the COVID-19 pandemic, the use of masks in daily life has become an important issue. The most important measure taken to prevent contagion is the use of masks. The aim of the study is to determine the effects of surgical masks used in every moment of life on physical performance in elderly individuals.

DETAILED DESCRIPTION:
Physical performance measurements were carried out by a physiotherapist using the Senior Fitness Test (SFT). Participants were informed about the procedure of the test. All participants performed two evaluation sessions by the SFT with and without using a surgical mask. The participants were randomly selected to perform the test whether with or without the surgical mask at first. The sessions were held at least 24 hours apart to prevent fatigue.

ELIGIBILITY:
Inclusion Criteria:

* geriatrics who had a score of ≥24 in the Mini Mental Test
* which evaluates the cognitive levels of individuals over the age of 65
* who were sufficient to perform physical function tests
* who had not been diagnosed with COVID-19 before

Exclusion Criteria:

* participants with severe respiratory disease (tuberculosis, severe COPD or bronchiectasis),
* uncontrolled cardiac arrhythmia, unstable angina, heart failure, severe kidney disease, neurological disorders that could cause consciousness change
* whose disease could not be controlled with medication

Ages: 65 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: Healthy individuals over the age of 65
Sampling Method: Non-Probability Sample
Enrollment: 46 (Actual)
Dates: Start 2020-09-10 (Actual); Primary Completion 2020-12-30 (Actual); Study Completion 2021-02-17 (Actual)

PRIMARY OUTCOMES:
Senior Fitness Test-Arm Curl | Baseline
  Upper extremity strength
Senior Fitness Test-Chair Stand Up and Sitting | Baseline
  Dynamic balance
Senior Fitness Test-Chair Sit and Reach | Baseline
  Lower extremity flexibility
Senior Fitness Test-Back Scratch | Baseline
  Upper extremity flexibility
Senior Fitness Test-Eight Foot Up and Go | Baseline
  Dynamic agility
Senior Fitness Test-Two-Minute Step Test | Baseline
  Aerobic endurance

CONTACTS AND LOCATIONS:
Overall Officials: Rıdvan Aktan, Study Chair — Izmir University of Economics; Özlem Akkoyun Sert, Study Chair — KTO Karatay University; Melike Akdam, Study Chair — KTO Karatay University; Buse Kılınç, Study Chair — KTO Karatay University; Sevgi Özalevli, Study Chair — Dokuz Eylul University
Locations (1):
- KTO Karatay University, Konya, Karatay, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No